CLINICAL TRIAL: NCT03913533
Title: Standard 6-sec Method Versus Tap-based Application Method to Assess Heart Rate at Birth - a Randomized Controlled Trial
Brief Title: Heart Rate Assessment at Birth Comparing Stethoscope Versus Tap-based Application
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding obtained
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro00089994
Record Dates: First submitted 2019-03-22; First posted 2019-04-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2021-09

CONDITIONS: Asphyxia Neonatorum; Birth Asphyxia
Keywords: Newborn; Heart rate assessment; Delivery Room
MeSH Terms: conditions — Asphyxia Neonatorum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: the outcome assessed will be masked to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Heart rate assessment using the Neonatal Resuscitation Program 6-sec assessment method At birth, the clinical team will place the stethoscope on the infant chest and calculate heart rate by listening to the heart beat for 6-sec and then compute the heart rate of the newborn infant.
  Interventions: Device: Heart rate assessment using the Neonatal Resuscitation Program 6-sec assessment method
- Intervention group (Experimental): Heart rate assessment using Tap-based smartphone application At birth, the clinical team will place the stethoscope on the infant chest and calculate heart rate using a Tap-based smartphone application by tapping the screen for 3 beats at that time a heart rate will be displayed.
  Interventions: Device: Heart rate assessment using Tap-based smartphone application

INTERVENTIONS:
Device: Heart rate assessment using the Neonatal Resuscitation Program 6-sec assessment method — Heart rate assessment using the Neonatal Resuscitation Program 6-sec assessment method At birth, the clinical team will place the stethoscope on the infant chest and calculate heart rate by listening to the heart beat for 6-sec and then compute the heart rate of the newborn infant.
  Arms: Control group
Device: Heart rate assessment using Tap-based smartphone application — At birth, the clinical team will place the stethoscope on the infant chest and calculate heart rate using a Tap-based smartphone application by tapping the screen for 3 beats at that time a heart rate will be displayed.
  Arms: Intervention group

SUMMARY:
Some newborn babies have difficulty breathing at birth and need help. When babies need help with breathing the clinical team, the team measures heart rate using a stethoscope to check its heart rate and figure out what kind of help they will need. If the heart rate is too low, the clinical team will begin to inflate the baby's lung. Knowing the baby's heart rate quickly is important but the stethoscope is inaccurate, and might delay start of resuscitation. Using a smartphone app that uses screen tapping with a stethoscope could allow heart rate to be measured much faster compared to the stethoscope and allow the clinical team to support the baby's needs better immediately after birth.

DETAILED DESCRIPTION:
Purpose

Nearly 10% of all infants born worldwide require respiratory support at birth and birth asphyxia remains one of the leading causes of infant morbidity and mortality. Neonatal resuscitation is the most effective strategy to deal with this condition. Moreover, an infant's heart rate (HR) is the most significant clinical parameter used to assess the need for and response to neonatal resuscitation. Currently, a newborn's HR is determined by auscultating or palpating of the umbilical cord. Although auscultation is more precise compared to palpation, both methods are inaccurate and tend to underestimate HR. The current resuscitation guidelines also recommend using electrocardiogram (ECG) and pulse oximetry, which allow for continuous monitoring, however are slow to apply and detect HR compared to stethoscopes. During neonatal resuscitation, an infant's HR is necessary to initiate resuscitation and to monitor the effectiveness of each intervention and therefore it becomes essential to accurately and quickly assess an infant's HR during this process. If HR is detected slowly or inaccurately, there is an increased risk that necessary interventions are not started or that certain interventions are prolonged, which could lead to increased morbidity and mortality of the infants. The recent advances in technology, namely the development of a smartphone tap application for HR assessment is promising as a novel tool for quick and accurate HR detection during neonatal resuscitation.

Hypothesis

The use of a tap-based smartphone application will be faster and more accurate when compared to standard auscultation with the 6-sec method to assess HR.

Justification

Simulation studies have shown that it is feasible to measure HR using a tap-based application. Moreover, the investigator's group has recently shown its reliability in an animal model of asphyxia-induced neonatal swine. The investigator showed its accuracy compared to the experimental gold standard carotid blood flow-derived HR assessments and report a median time of 3 sec for assessment, which is less than the current recommended time for auscultation. However, no study has been performed in the delivery room in newborn babies at birth. Therefore, the investigator aim to compare the tap-based application to the current 6-sec standard approach to assess HR during neonatal resuscitation in the delivery room. Ehe investigator anticipate this study will allow us to determine the most reliable approach for initial assessment to reduce neonatal morbidity and mortality outcomes.

Objectives

To examine (i) accuracy and (ii) speed to assess HR using auscultation with a tap-based application during neonatal resuscitation.

Research Method/Procedures

The proposed study is a randomized controlled trial comparing two different approaches to accurately assess HR. The investigator will compare the routinely used Neonatal Resuscitation Program 6-sec method with a stethoscope using two different methods of auscultation [6-sec method and tap-based method (NeoTapLS, Tap4Life, Stockholm, Sweden)] to accurately assess HR immediately after birth. The investigator aim to collect the data over a period of 12 months.

Two investigators in addition to the clinical team will attend the delivery of newborn infants. Immediately after birth the infant will be placed on a resuscitation trolley where a pulse oximeter will be attached to the right hand. At the same time three ECG leads will be placed on the infant's chest. Simultaneously the stethoscope will be placed by one of the investigators on the infants' chest to obtain the HR . In the alternative setup, stethoscope will be used in combination with the tap-based application.

In both setups, the time needed to display a HR will be recorded for all devices. All infants will have routine HR measured using ECG, which will be used as comparison for accuracy

ELIGIBILITY:
Inclusion Criteria:

* All newborn infants delivered in the Royal Alexandra Hospital (RAH) 22+0-41+6 weeks gestation.

Exclusion Criteria:

* Infants will be excluded if parents refused to consent to the study.

Max Age: 5 Minutes | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-12-16 (Actual); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to obtain Heart rate | within the first 60 seconds form birth
  Time to obtain Heart rate form birth

SECONDARY OUTCOMES:
Accuracy of heart rate assessment using either technique | within the first 60 seconds form birth
  Accuracy of heart rate assessment using tap-based application or 6-sec method

CONTACTS AND LOCATIONS:
Overall Officials: Georg Schmolzer, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- Royal Alexandra Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
requests can be made to the PI
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: once study is completed and published
Access Criteria: email requests to the PI

REFERENCES:
- [Result] Saugstad OD, Ramji S, Rootwelt T, Vento M. Response to resuscitation of the newborn: early prognostic variables. Acta Paediatr. 2005 Jul;94(7):890-5. doi: 10.1111/j.1651-2227.2005.tb02007.x. PMID 16188811
- [Result] Wyckoff MH, Aziz K, Escobedo MB, Kapadia VS, Kattwinkel J, Perlman JM, Simon WM, Weiner GM, Zaichkin JG. Part 13: Neonatal Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S543-60. doi: 10.1161/CIR.0000000000000267. No abstract available. PMID 26473001
- [Result] Duryea EL, Nelson DB, Wyckoff MH, Grant EN, Tao W, Sadana N, Chalak LF, McIntire DD, Leveno KJ. The impact of ambient operating room temperature on neonatal and maternal hypothermia and associated morbidities: a randomized controlled trial. Am J Obstet Gynecol. 2016 Apr;214(4):505.e1-505.e7. doi: 10.1016/j.ajog.2016.01.190. Epub 2016 Feb 10. PMID 26874298
- [Result] Kamlin CO, O'Donnell CP, Everest NJ, Davis PG, Morley CJ. Accuracy of clinical assessment of infant heart rate in the delivery room. Resuscitation. 2006 Dec;71(3):319-21. doi: 10.1016/j.resuscitation.2006.04.015. Epub 2006 Sep 20. PMID 16989935
- [Result] Kamlin CO, Dawson JA, O'Donnell CP, Morley CJ, Donath SM, Sekhon J, Davis PG. Accuracy of pulse oximetry measurement of heart rate of newborn infants in the delivery room. J Pediatr. 2008 Jun;152(6):756-60. doi: 10.1016/j.jpeds.2008.01.002. Epub 2008 Mar 6. PMID 18492509
- [Result] Kopotic RJ, Lindner W. Assessing high-risk infants in the delivery room with pulse oximetry. Anesth Analg. 2002 Jan;94(1 Suppl):S31-6. PMID 11900034
- [Result] Luong DH, Cheung PY, O'Reilly M, Lee TF, Schmolzer GM. Electrocardiography vs. Auscultation to Assess Heart Rate During Cardiac Arrest With Pulseless Electrical Activity in Newborn Infants. Front Pediatr. 2018 Nov 27;6:366. doi: 10.3389/fped.2018.00366. eCollection 2018. PMID 30538976
- [Result] Patel S, Cheung PY, Solevag AL, Barrington KJ, Kamlin COF, Davis PG, Schmolzer GM. Pulseless electrical activity: a misdiagnosed entity during asphyxia in newborn infants? Arch Dis Child Fetal Neonatal Ed. 2019 Mar;104(2):F215-F217. doi: 10.1136/archdischild-2018-314907. Epub 2018 Jun 12. PMID 29895572
- [Result] Owen CJ, Wyllie JP. Determination of heart rate in the baby at birth. Resuscitation. 2004 Feb;60(2):213-7. doi: 10.1016/j.resuscitation.2003.10.002. PMID 15036740
- [Result] Voogdt KG, Morrison AC, Wood FE, van Elburg RM, Wyllie JP. A randomised, simulated study assessing auscultation of heart rate at birth. Resuscitation. 2010 Aug;81(8):1000-3. doi: 10.1016/j.resuscitation.2010.03.021. Epub 2010 May 18. PMID 20483522
- [Result] Binotti M, Cavallin F, Ingrassia PL, Pejovic NJ, Monzani A, Genoni G, Trevisanuto D. Heart rate assessment using NeoTapAdvancedSupport: a simulation study. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F440-F442. doi: 10.1136/archdischild-2018-315408. Epub 2018 Sep 27. PMID 30262463